CLINICAL TRIAL: NCT02634411
Title: Impact of the Duration of Antibiotics on Clinical Events in Patients With Pseudomonas Aeruginosa Ventilator-associated Pneumonia : a Randomized Controlled Study (iDIAPASON)
Brief Title: Impact of the Duration of Antibiotics on Clinical Events in Patients With Pseudomonas Aeruginosa Ventilator-associated Pneumonia (iDIAPASON)
Acronym: iDIAPASON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 140923; AOM 14515 (Other: AOM); IDRCB n°: 2015-A00375-44 (Other: IDRCP)
Record Dates: First submitted 2015-11-19; First posted 2015-12-18 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Ventilator Associated; Pneumonia; Antibiotic treatment; Pseudomonas aeruginosa
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia; Pseudomonas Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8 days of effective antibiotic treatment (Experimental): Antibiotic treatment should be started just after realization of bacteriological sampling, and then converted into a narrow-spectrum therapy, based on culture results, for a total duration of effective antibiotic therapy against PA of 8 days.
  Interventions: Drug: 8 days of effective antibiotic treatment
- 15 days of effective antibiotic treatment (Sham Comparator): Antibiotic treatment should be started just after realization of bacteriological sampling, and then converted into a narrow-spectrum therapy, based on culture results, for a total duration of effective antibiotic therapy against PA of 15 days.
  Interventions: Drug: 15 days of effective antibiotic treatment

INTERVENTIONS:
Drug: 8 days of effective antibiotic treatment — Antibiotics used for usual care in PA-VAP treatment : Penicillins, Cephalosporins, Monobactams, Carbapenems, Fluoroquinolones, Aminoglycosides (list not exhaustive).
  Antibiotic treatment should be started just after realization of bacteriological sampling, and then converted into a narrow-spectrum therapy, based on culture results, for a total duration of effective antibiotic therapy against pseudomona aeruginosa of 8 days.
  Arms: 8 days of effective antibiotic treatment
Drug: 15 days of effective antibiotic treatment — Antibiotics used for usual care in PA-VAP treatment : Penicillins, Cephalosporins, Monobactams, Carbapenems, Fluoroquinolones, Aminoglycosides (list not exhaustive).
  Antibiotic treatment should be started just after realization of bacteriological sampling, and then converted into a narrow-spectrum therapy, based on culture results, for a total duration of effective antibiotic therapy against pseudomona aeruginosa of 15 days.
  Arms: 15 days of effective antibiotic treatment

SUMMARY:
Ventilator-associated pneumonia (VAP) accounts for 25% of infections in intensive care units (Réseau RAISIN 2012). A short duration (8 days; SD) vs. long duration (15 days; LD) of antibiotic therapy has a comparable clinical efficacy with less antibiotic use and less multidrug-resistant pathogens (MDR) emergence. These results have led the American Thoracic Society to recommend SD therapy for VAP, with the exception of documented VAP of non-fermenting Gram negative bacilli (NF-GNB), including Pseudomonas aeruginosa (PA-VAP), due to the absence of studies focusing specifically on PA-VAP. Thus the beneficial effect of SD therapy in PA-VAP is still a matter of debate. In a small (n=127) subgroup analysis, a higher rate of recurrence with SD therapy (n=21, 32.8%) has been observed compared with LD therapy group (n=12, 19.0%). Unfortunately, the definition of recurrence was essentially based on microbiological rather than clinical data, and the higher rate of recurrence observed could rather reflect a higher rate of colonization more than a new infection.

Interestingly, a trend for a lower rate of mortality was also observed in the SD group (n=15, 23.4%) compared with the LD group (n=19, 30.2%), but this study was clearly underpowered to detect a difference of mortality between groups.

The two strategies were considered as not different, for the risk of mortality in a recent meta-analysis, performed on the very few available studies (n=2), that (OR = 1.33, 95% CI [0.33 to 5.26] for SD vs. LD strategies respectively). However, this conclusion remains questionable considering the large confidence interval of the risk and the power of these studies.

Primary objective and assessment criterion: To assess the non-inferiority of a short duration of antibiotics (8 days) vs. prolonged antibiotic therapy (15 days) in P. aeruginosa ventilator-associated pneumonia (PA-VAP) on a composite end-point combining Day-90 mortality and PA-VAP recurrence rate during hospitalization in the ICU.

Study Design :

Randomized, open-labeled non inferiority controlled trial 32 French Intensive Care Units participating to the study

Research period:

Total study duration: 27 months Inclusion period: 24 months Duration of participation for a patient: 90 days

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a major cause of morbidity and mortality in the ICU, accounting for 25% of infections in intensive care units (Réseau RAISIN 2012). From 1975 to 2003, the incidence of hospital-acquired pneumonia caused by Pseudomonas aeruginosa (PA) has almost doubled, from 9.6% to 18.1%. In a US national large-scale survey, PA was the most frequently isolated gram-negative aerobic bacterium from ICUs (23%) and also the most frequent bacterium isolated from the respiratory tract (31.6%).

PA-VAP is associated with a high mortality ranging from 40% up to 69%, and with high rates of recurrence despite adequate antimicrobial therapy. In a large randomized trial regarding the optimal duration of antibiotic therapy in overall VAPs, the rate of recurrence among the subgroup of non-fermenting Gram negative bacilli (NF-GNB) documented VAP varied between 19.0% and 32.8%, according to the randomization arm. Finally, a recently published cohort about 393 PA-VAP in 314 patients, the composite criteria failure treatment (death and recurrence) occured in 112 cases (28.5%).

Hypothesis A short duration antibiotherapy (8 days) vs. long duration antibiotherapy (15 days) in treatment of Pseudomonas aeruginosa Ventilator-Associated Pneumonia (PA-VAP) is safe and not associated with an increased mortality or recurrence rate of PA-VAP.

The demonstration of this hypothesis could lead to decrease antibiotic exposure during the hospitalization in the Intensive Care Unit (ICU) and in turn reduce the acquisition and the spread of multidrug-resistant pathogens (MDR).

Objectives

1. Primary objective To assess the non-inferiority of a short duration of antibiotics (8 days) vs. prolonged antibiotic therapy (15 days) in Pseudomonas aeruginosa ventilator-associated pneumonia (PA-VAP) on morbi-mortality at 90 days.
2. Secondary objectives

To compare between short and long duration of antibiotics on:

* mortality in the ICU
* morbidity in the ICU (mechanical ventilation, duration of hospitalization)
* exposure and acquisition of MDR during hospitalization
* number and types of extrapulmonary infections

Plan for the research

1. Concise description of the primary and secondary assessment criteria

   - Primary assessment criterion: A composite endpoint combining Day-90 mortality and PA-VAP recurrence rate during hospitalization in the ICU (within 90 days).

   Recurrence will be defined a posteriori by 3 independent experts with predefined criteria: clinical suspicion of VAP (≥ two criteria including: fever> 38.5°C, leukocytosis > 10 Giga/L or leukopenia < 4 Giga/L, purulent tracheobronchial secretions and a new or persistent infiltrate on chest radiography). associated with a positive quantitative culture of a respiratory sample (bronchoalveolar lavage fluid (significant threshold ≥104 colony-forming units/mL) or plugged telescopic catheter (significant threshold ≥103 colony-forming units/mL) or quantitative endotracheal aspirate distal pulmonary secretion samples (significant threshold ≥106 colony-forming units/mL)).
   * Secondary assessment criteria:

     1. D30 and D90 mortality rate (%)
     2. Morbidity by:

        Duration of mechanical ventilation (days) Duration of hospitalization in ICU (days)
     3. Exposure to antibiotics during the hospitalization in the ICU (days)
     4. Number and types of extrapulmonary infections during the hospitalization in the ICU (n)
     5. Acquisition of MDR during the hospitalization in the ICU (swab sample of rectum and anterior nares)
2. Description of research methodology

Randomized, open-labeled non inferiority trial comparing to parallel groups:

* 8 days of antibiotic therapy
* 15 days of antibiotic therapy

Antibiotic therapy Antibiotic treatment should be started just after realization of bacteriological sampling, without waiting for the result. The choice of initial antibiotic therapy will be left to the discretion of the physician but will be essentially based on the clinical context, previously antibiotic therapy, the presence or absence of risk factors for MDR (antibiotics or hospitalization in previous 90 days, current hospitalization ≥ 5 days, MV ≥ 5 days, supported in a dialysis center or residency in a nursing home), local epidemiological data, and finally if the patient is already known as being colonized by a MDR. Investigators would be strongly encouraged to convert this initial regimen into a narrow- spectrum therapy, based on culture results.

All antibiotics would be withdrawn, either at the end of day 8 or day 15, according to the randomization assignment, except those prescribed for a documented pulmonary infection recurrence before that day.

An algorithm for the initial prescription of antibiotics will be established in each ICU, the algorithm will be adapted whenever necessary to changes in the local ecology.

Number of centres participating 42 french Intensive Care Units (ICUs)

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Mechanical ventilation ≥ 48 hours
* Documented Pseudomonas aeruginosa ventilator-associated pneumonia:

  * Clinical suspicion (≥ two criteria including: fever> 38.5°C,leukocytosis > 10 Giga/L or leukopenia < 4 Giga/L, purulent tracheobronchial secretions and a new or persistent infiltrate on chest radiography).
  * Documented Pseudomonas aeruginosa positive quantitative culture of a respiratory sample: bronchoalveolar lavage fluid (significant threshold, >104cfu/ml) or plugged telescopic catheter (significant threshold, >103cfu/ml) or quantitative endotracheal aspirate (significant threshold, >106cfu/ml).
* Written informed consent
* Patient affiliated to French social security

Exclusion Criteria:

* Immunocompromised patients (HIV, immunosuppressive therapy, corticosteroids> 0.5 mg / kg per day for more than a month)
* Patients receiving antibiotic therapy for extrapulmonary infection
* Patients in whom a procedure of withdrawing life-sustaining treatment has been established
* Pregnancy
* Patients included in another interventional study
* Chronic pulmonary colonization with Pseudomonas aeruginosa: patients with Chronic Obstructive Pulmonary Disease (COPD) or bronchiectasis, with a positive respiratory sample at infra threshold rate for Pseudomonas aeruginosa (ie<103 CFUs/mL for protected specimen brush or <106 CFUs/mL for tracheal aspirate), obtained in the absence of pneumonia or exacerbation during the 6 months before the ICU admission.
* Patient under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
A composite endpoint of morbi-mortality combining Day-90 mortality and PA-VAP recurrence rate during hospitalization in the ICU (within 90 days). | 90 days after effective antibiotherapy
  A composite endpoint combining Day-90 mortality and PA-VAP recurrence rate during hospitalization in the ICU (within 90 days).
  Recurrence will be defined a posteriori by 3 independent experts with predefined criteria: clinical suspicion of VAP (≥ two criteria including: fever> 38.5 ° C, leukocytosis > 10 Giga/L or leukopenia < 4 Giga/L, purulent tracheobronchial secretions and a new or persistent infiltrate on chest radiography) associated with a positive quantitative culture of a respiratory sample (bronchoalveolar lavage fluid (significant threshold ≥104 colony-forming units/mL) or plugged telescopic catheter (significant threshold ≥103 colony-forming units/mL) or quantitative endotracheal aspirate distal pulmonary secretion samples (significant threshold ≥106 colony-forming units/mL)).

SECONDARY OUTCOMES:
Measure of mortality rate (%) in the ICU | Day 30 and Day 90 after effective antibiotherapy
Measure of morbidity in ICU by duration of mechanical ventilation (days) | Day 30 and Day 90 after effective antibiotherapy
Measure of morbidity in ICU by duration of hospitalization in ICU (days) | Day 30 and Day 90 after effective antibiotherapy
Acquisition of MDR during the hospitalization in the ICU. | during stay in the ICU : up to 90 days
Exposure to antibiotics during the hospitalization in the ICU (days) | during stay in the ICU : up to 90 days
Number of extrapulmonary infections during the hospitalization in the ICU | during stay in the ICU : up to 90 days
Type of extrapulmonary infections during the hospitalization in the ICU | during stay in the ICU : up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Bouglé, MD, Principal Investigator — APHP
Locations (1):
- Anesthesiology and Critical Care Medicine Institut de Cardiologie, Groupe Hospitalier Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Background] Gaynes R, Edwards JR; National Nosocomial Infections Surveillance System. Overview of nosocomial infections caused by gram-negative bacilli. Clin Infect Dis. 2005 Sep 15;41(6):848-54. doi: 10.1086/432803. Epub 2005 Aug 16. PMID 16107985
- [Background] Neuhauser MM, Weinstein RA, Rydman R, Danziger LH, Karam G, Quinn JP. Antibiotic resistance among gram-negative bacilli in US intensive care units: implications for fluoroquinolone use. JAMA. 2003 Feb 19;289(7):885-8. doi: 10.1001/jama.289.7.885. PMID 12588273
- [Background] Crouch Brewer S, Wunderink RG, Jones CB, Leeper KV Jr. Ventilator-associated pneumonia due to Pseudomonas aeruginosa. Chest. 1996 Apr;109(4):1019-29. doi: 10.1378/chest.109.4.1019. PMID 8635325
- [Background] Trouillet JL, Vuagnat A, Combes A, Kassis N, Chastre J, Gibert C. Pseudomonas aeruginosa ventilator-associated pneumonia: comparison of episodes due to piperacillin-resistant versus piperacillin-susceptible organisms. Clin Infect Dis. 2002 Apr 15;34(8):1047-54. doi: 10.1086/339488. Epub 2002 Mar 15. PMID 11914992
- [Background] Garnacho-Montero J, Sa-Borges M, Sole-Violan J, Barcenilla F, Escoresca-Ortega A, Ochoa M, Cayuela A, Rello J. Optimal management therapy for Pseudomonas aeruginosa ventilator-associated pneumonia: an observational, multicenter study comparing monotherapy with combination antibiotic therapy. Crit Care Med. 2007 Aug;35(8):1888-95. doi: 10.1097/01.CCM.0000275389.31974.22. PMID 17581492
- [Background] Planquette B, Timsit JF, Misset BY, Schwebel C, Azoulay E, Adrie C, Vesin A, Jamali S, Zahar JR, Allaouchiche B, Souweine B, Darmon M, Dumenil AS, Goldgran-Toledano D, Mourvillier BH, Bedos JP; OUTCOMEREA Study Group. Pseudomonas aeruginosa ventilator-associated pneumonia. predictive factors of treatment failure. Am J Respir Crit Care Med. 2013 Jul 1;188(1):69-76. doi: 10.1164/rccm.201210-1897OC. PMID 23641973
- [Background] Chastre J, Wolff M, Fagon JY, Chevret S, Thomas F, Wermert D, Clementi E, Gonzalez J, Jusserand D, Asfar P, Perrin D, Fieux F, Aubas S; PneumA Trial Group. Comparison of 8 vs 15 days of antibiotic therapy for ventilator-associated pneumonia in adults: a randomized trial. JAMA. 2003 Nov 19;290(19):2588-98. doi: 10.1001/jama.290.19.2588. PMID 14625336
- [Background] Klompas M. Does this patient have ventilator-associated pneumonia? JAMA. 2007 Apr 11;297(14):1583-93. doi: 10.1001/jama.297.14.1583. PMID 17426278
- [Background] Pugin J, Auckenthaler R, Mili N, Janssens JP, Lew PD, Suter PM. Diagnosis of ventilator-associated pneumonia by bacteriologic analysis of bronchoscopic and nonbronchoscopic "blind" bronchoalveolar lavage fluid. Am Rev Respir Dis. 1991 May;143(5 Pt 1):1121-9. doi: 10.1164/ajrccm/143.5_Pt_1.1121. PMID 2024824
- [Background] Johanson WG Jr, Pierce AK, Sanford JP, Thomas GD. Nosocomial respiratory infections with gram-negative bacilli. The significance of colonization of the respiratory tract. Ann Intern Med. 1972 Nov;77(5):701-6. doi: 10.7326/0003-4819-77-5-701. No abstract available. PMID 5081492
- [Background] Baram D, Hulse G, Palmer LB. Stable patients receiving prolonged mechanical ventilation have a high alveolar burden of bacteria. Chest. 2005 Apr;127(4):1353-7. doi: 10.1378/chest.127.4.1353. PMID 15821215
- [Background] El Solh AA, Akinnusi ME, Wiener-Kronish JP, Lynch SV, Pineda LA, Szarpa K. Persistent infection with Pseudomonas aeruginosa in ventilator-associated pneumonia. Am J Respir Crit Care Med. 2008 Sep 1;178(5):513-9. doi: 10.1164/rccm.200802-239OC. Epub 2008 May 8. PMID 18467510
- [Background] Borg MA. Bed occupancy and overcrowding as determinant factors in the incidence of MRSA infections within general ward settings. J Hosp Infect. 2003 Aug;54(4):316-8. doi: 10.1016/s0195-6701(03)00153-1. PMID 12919764
- [Background] Trouillet JL, Chastre J, Vuagnat A, Joly-Guillou ML, Combaux D, Dombret MC, Gibert C. Ventilator-associated pneumonia caused by potentially drug-resistant bacteria. Am J Respir Crit Care Med. 1998 Feb;157(2):531-9. doi: 10.1164/ajrccm.157.2.9705064. PMID 9476869
- [Background] Micek ST, Ward S, Fraser VJ, Kollef MH. A randomized controlled trial of an antibiotic discontinuation policy for clinically suspected ventilator-associated pneumonia. Chest. 2004 May;125(5):1791-9. doi: 10.1378/chest.125.5.1791. PMID 15136392
- [Background] Kollef MH, Kollef KE. Antibiotic utilization and outcomes for patients with clinically suspected ventilator-associated pneumonia and negative quantitative BAL culture results. Chest. 2005 Oct;128(4):2706-13. doi: 10.1378/chest.128.4.2706. PMID 16236946
- [Background] Pugh R, Grant C, Cooke RP, Dempsey G. Short-course versus prolonged-course antibiotic therapy for hospital-acquired pneumonia in critically ill adults. Cochrane Database Syst Rev. 2011 Oct 5;(10):CD007577. doi: 10.1002/14651858.CD007577.pub2. PMID 21975771
- [Background] Bouadma L, Luyt CE, Tubach F, Cracco C, Alvarez A, Schwebel C, Schortgen F, Lasocki S, Veber B, Dehoux M, Bernard M, Pasquet B, Regnier B, Brun-Buisson C, Chastre J, Wolff M; PRORATA trial group. Use of procalcitonin to reduce patients' exposure to antibiotics in intensive care units (PRORATA trial): a multicentre randomised controlled trial. Lancet. 2010 Feb 6;375(9713):463-74. doi: 10.1016/S0140-6736(09)61879-1. Epub 2010 Jan 25. PMID 20097417
- [Background] Stolz D, Smyrnios N, Eggimann P, Pargger H, Thakkar N, Siegemund M, Marsch S, Azzola A, Rakic J, Mueller B, Tamm M. Procalcitonin for reduced antibiotic exposure in ventilator-associated pneumonia: a randomised study. Eur Respir J. 2009 Dec;34(6):1364-75. doi: 10.1183/09031936.00053209. Epub 2009 Sep 24. PMID 19797133
- [Background] Amour J, Birenbaum A, Langeron O, Le Manach Y, Bertrand M, Coriat P, Riou B, Bernard M, Hausfater P. Influence of renal dysfunction on the accuracy of procalcitonin for the diagnosis of postoperative infection after vascular surgery. Crit Care Med. 2008 Apr;36(4):1147-54. doi: 10.1097/CCM.0b013e3181692966. PMID 18379240
- [Background] Schuetz P, Albrich W, Christ-Crain M, Chastre J, Mueller B. Procalcitonin for guidance of antibiotic therapy. Expert Rev Anti Infect Ther. 2010 May;8(5):575-87. doi: 10.1586/eri.10.25. PMID 20455686
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Fekih Hassen M, Ayed S, Ben Sik Ali H, Gharbi R, Marghli S, Elatrous S. [Duration of antibiotic therapy for ventilator-associated pneumonia: comparison of 7 and 10 days. A pilot study]. Ann Fr Anesth Reanim. 2009 Jan;28(1):16-23. doi: 10.1016/j.annfar.2008.10.021. Epub 2008 Dec 18. French. PMID 19097848
- [Background] Capellier G, Mockly H, Charpentier C, Annane D, Blasco G, Desmettre T, Roch A, Faisy C, Cousson J, Limat S, Mercier M, Papazian L. Early-onset ventilator-associated pneumonia in adults randomized clinical trial: comparison of 8 versus 15 days of antibiotic treatment. PLoS One. 2012;7(8):e41290. doi: 10.1371/journal.pone.0041290. Epub 2012 Aug 31. PMID 22952580
- [Background] Kollef MH, Chastre J, Clavel M, Restrepo MI, Michiels B, Kaniga K, Cirillo I, Kimko H, Redman R. A randomized trial of 7-day doripenem versus 10-day imipenem-cilastatin for ventilator-associated pneumonia. Crit Care. 2012 Nov 13;16(6):R218. doi: 10.1186/cc11862. PMID 23148736
- [Background] Dimopoulos G, Poulakou G, Pneumatikos IA, Armaganidis A, Kollef MH, Matthaiou DK. Short- vs long-duration antibiotic regimens for ventilator-associated pneumonia: a systematic review and meta-analysis. Chest. 2013 Dec;144(6):1759-1767. doi: 10.1378/chest.13-0076. PMID 23788274
- [Background] Hanberger H, Garcia-Rodriguez JA, Gobernado M, Goossens H, Nilsson LE, Struelens MJ. Antibiotic susceptibility among aerobic gram-negative bacilli in intensive care units in 5 European countries. French and Portuguese ICU Study Groups. JAMA. 1999 Jan 6;281(1):67-71. doi: 10.1001/jama.281.1.67. PMID 9892453
- [Background] Cosgrove SE. The relationship between antimicrobial resistance and patient outcomes: mortality, length of hospital stay, and health care costs. Clin Infect Dis. 2006 Jan 15;42 Suppl 2:S82-9. doi: 10.1086/499406. PMID 16355321
- [Background] Paterson DL. The epidemiological profile of infections with multidrug-resistant Pseudomonas aeruginosa and Acinetobacter species. Clin Infect Dis. 2006 Sep 1;43 Suppl 2:S43-8. doi: 10.1086/504476. PMID 16894514
- [Background] Kalfon P, Giraudeau B, Ichai C, Guerrini A, Brechot N, Cinotti R, Dequin PF, Riu-Poulenc B, Montravers P, Annane D, Dupont H, Sorine M, Riou B; CGAO-REA Study Group. Tight computerized versus conventional glucose control in the ICU: a randomized controlled trial. Intensive Care Med. 2014 Feb;40(2):171-181. doi: 10.1007/s00134-013-3189-0. Epub 2014 Jan 14. PMID 24420499
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006
- [Background] Dunnett CW, Gent M. Significance testing to establish equivalence between treatments, with special reference to data in the form of 2X2 tables. Biometrics. 1977 Dec;33(4):593-602. PMID 588654
- [Background] Le Gall JR, Lemeshow S, Saulnier F. A new Simplified Acute Physiology Score (SAPS II) based on a European/North American multicenter study. JAMA. 1993 Dec 22-29;270(24):2957-63. doi: 10.1001/jama.270.24.2957. PMID 8254858
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Derived] Foucrier A, Dessalle T, Tuffet S, Federici L, Dahyot-Fizelier C, Barbier F, Pottecher J, Monsel A, Hissem T, Lefrant JY, Demoule A, Constantin JM, Rousseau A, Simon T, Leone M, Bougle A; iDIAPASON Trial Investigators. Association between combination antibiotic therapy as opposed as monotherapy and outcomes of ICU patients with Pseudomonas aeruginosa ventilator-associated pneumonia: an ancillary study of the iDIAPASON trial. Crit Care. 2023 May 30;27(1):211. doi: 10.1186/s13054-023-04457-y. PMID 37254209
- [Derived] Bougle A, Foucrier A, Dupont H, Montravers P, Ouattara A, Kalfon P, Squara P, Simon T, Amour J; iDIAPASON study group. Impact of the duration of antibiotics on clinical events in patients with Pseudomonas aeruginosa ventilator-associated pneumonia: study protocol for a randomized controlled study. Trials. 2017 Jan 23;18(1):37. doi: 10.1186/s13063-017-1780-3. PMID 28114979